CLINICAL TRIAL: NCT03960723
Title: Descriptive Study to Evaluate the Understanding Degree of Informed Consent in Surgical Procedures
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CIP-2019-25
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Informed Consent
Keywords: Informed consent
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A questionnaire asking the patients for several questions related to the Informed Consent Form they have signed before surgery, will be administered.

SUMMARY:
The Informed Consent (IC) of a medical procedure is the aceptation of a diagnostic or therapeutic procedure by the patient, after receiving the necessary and accurate information about it. Freedom, information and understanding have to be the main requirements in this proccess.

The main goal of this study is to assess if patients that are going to be operated at Hospital de la Santa Creu i Sant Pau in the CSI (Surgery without previous hospitalization) unit, really understood the information about the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery and admitted by CSI unit
* Provide written informed consent to participate in the study

Exclusion Criteria:

* Patients who need a legal representative to read, understand and sign the CI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years, who undergoing surgery and are admitted by CSI unit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Understanding degree | Before procedure
  Assessment of the understanding degree of the IC by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Mª Antonijoan Arbos, MD, PhD, Principal Investigator — Institut de Recerca de l´Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain